CLINICAL TRIAL: NCT04415567
Title: Adjuvant Lenvatinib Prevents Recurrence of High-risk Patients With Hepatitis B Virus-related Hepatocellular Carcinoma Following Liver Transplantation: a Retrospective Case Control Study
Brief Title: Adjuvant Lenvatinib Prevents Recurrence of High-risk Patients With HBV-related HCC After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Jinyang Gu (Other)
Responsible Party: Sponsor-Investigator, Jinyang Gu, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: XH-20-010
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; liver transplantation; lenvatinib; adjuvant therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- lenvatinib: high-risk patients with HBV-related HCC who took lenvatinib as adjuvant therapy after liver transplantation
  Interventions: Drug: Lenvatinib
- control: high-risk patients with HBV-related HCC who received routine treatment and follow-up after liver transplantation

INTERVENTIONS:
Drug: Lenvatinib — The patients in lenvatinib group received oral lenvatinib (Eisai, Japan) 12 mg/day (for bodyweight (BW) ≥60 kg) or 8 mg/day (for BW <60 kg) in 28-day cycles until HCC recurrence or serious adverse events (SAEs) or voluntary withdrawal. Dose interruptions followed by reductions for lenvatinib-related toxicities (to 8 mg and 4 mg/day, or 4 mg every other day) were permitted. All 14 patients took lenvatinib for more than 3 cycles.
  Groups: lenvatinib

SUMMARY:
High-risk patients with hepatitis B virus (HBV)-related hepatocellular carcinoma (HCC) suffer from a high ratio of recurrence after liver transplantation (LT). Lenvatinib, as a novel targeted drug, has shown an excellent effect in the treatment of advanced HCC, but there is no study on its effect in preventing HCC recurrence in the patients undergoing transplantation. Therefore, to evaluate the role of adjuvant lenvatinib in preventing recurrence of high-risk LT recipients with HBV-related HCC, the investigators retrospectively analyzed 23 high-risk patients consisting of lenvatinib group (n=14) and control group (n=9) with HBV-related HCC who underwent LT. Disease-free survival (DFS) and HCC recurrence of the two groups were compared. The adverse events (AEs) and drug tolerance of lenvatinib were evaluated.

DETAILED DESCRIPTION:
The investigators retrospectively reviewed 23 Chinese HCC patients with HBV infection, who underwent LT in our hospital from June 2018 to December 2019. All donor grafts were allocated by the China Organ Transplant Response System. All these patients were diagnosed by histology and were defined as "high-risk" for recurrence.

The participants were divided into lenvatinib group and control group according to their willingness to take lenvatinib as adjuvant therapy after LT. Of the 23 patients, 14 pantients in lenvatinib group began to take lenvatinib about a month after LT except for routine treatment, while the other 9 patients in control group received routine treatment and follow-up after transplantation. Clinical data and demographic characteristics was obtained. This study was conducted according to the 1975 Declaration of Helsinki and approved by Ethics Committee of Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine (No. XHEC-D-2020-068). All patients enrolled in this study provided informed consent.

Usage of lenvatinib and immunosuppressants The participants in lenvatinib group received oral lenvatinib (Eisai, Japan) 12 mg/day (for bodyweight (BW) ≥60 kg) or 8 mg/day (for BW <60 kg) in 28-day cycles until HCC recurrence or serious adverse events (SAEs) or voluntary withdrawal. Dose interruptions followed by reductions for lenvatinib-related toxicities (to 8 mg and 4 mg/day, or 4 mg every other day) were permitted. All 14 patients took lenvatinib for more than 3 cycles.

The induction immunosuppression strategies for all participants enrolled in the study involved IV infusion of 20mg of basiliximab within 2 hours prior to operation and a second dose 4 days later, oral tacrolimus started on the fourth day after LT at a dose of 0.04mg/kg (BW) and adjusted according to its plasma concentration, taking mycophenolate mofetil (MMF) from the next day after surgery at a dose of 500mg/kg(BW), and rapid withdrawal of glucocorticoids with the initial dose of 500mg. Maintenance immunosuppression which was started about one month after LT included sirolimus (4 mg/M2 per day) plus oral tacrolimus with the plasma concentration maintained at 5-8 ng/ml.

All patients were followed up monthly within six months after LT and every three months within two years. During each follow-up, complete blood count, urinalysis, serum AFP level, liver and kidney function test, and blood concentration of FK506 were recorded. Chest and abdominal computed tomography was implemented at 3 months, 6 months, 12 months, and annually thereafter. Other radiological examinations such as radionuclide bone scan, magnetic resonance imaging (MRI) and positron emission tomography (PET) were obtained when local recurrence or distant metastasis was suspected.

The DFS was defined as the period between the day of LT and the day of HCC recurrence confirmed by imaging, while the OS was defined as the duration from LT to death of patients for any reason or to end of follow-up. Common terminology criteria for adverse events version 5.0 (CTCAE V5.0) was used to assess the AE during oral administration of lenvatinib. The FK506 dosage and blood concentration of each patients in the first six months after liver LT was recorded for evaluate the influence of lenvatinib on the immunosuppressive therapy.

Mean and standard deviations were used for descriptive statistics. The patient characteristics in each group were compared by one-way ANOVA and chi-square tests. Repeated measures analysis of variances was used for comparing the difference of FK506 dosage and blood concentration between two groups. The OS and DFS were statistically analyzed by the Kaplan-Meier method. Statistical significance was set at P<0.05. All statistical analyses were performed using SPSS software Version 10.0.

ELIGIBILITY:
Inclusion Criteria:

1. The recipients who underwent liver transplantation with the pathologic diagnosis of hepatocellular carcinoma.
2. The extrahepatic metastasis was excluded preoperatively.
3. The patients were defined as "high-risk" for recurrence according to the following criteria:

(1) beyond Milan criteria confirmed either by radiology before LT or by pathology after LT, (2) tumor with intrahepatic vascular invasion, (3) Alpha-fetoprotein (AFP)≥400ng/L before LT, (4) presence of microvascular invasion (MVI), (5) tumor with histological poor differentiation according to Edmondson-Steiner classification system(21), (6) multiple satellite lesions around the largest tumors detected either by radiology before LT or by histology after LT, (7) tumor penetrating hepatic capsule, (8) recurrent HCC after resection. 4. ECOG score between 0-1 within 1 week before took lenvatinib. 5. The patients have received regular antiviral treatment. 6. Life expectancy more than 3 months.

Exclusion Criteria:

1. The patients took lenvatinib before liver transplantation and assessed as SD or PD according to the mRECIST criteria.
2. The patients suffered from other incurable malignancies within 5 years or at the same time.
3. Distant metastasis of tumor was confirmed by imaging before or within 1 month after transplantation.
4. The patients have not received regular antiviral treatment.
5. The patients had a history of mental illness or abuse of psychoactive drugs.
6. The patients deemed unsuitable by attending doctors.

Ages: 8 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohorts in the study involved the patients who underwent liver transplantation for HBV-related HCC and were diagnosed as "high-risk" for recurrence according the above criteria.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | up to 3 years
  The disease-free survival (DFS) was defined as the period between the day of LT and the day of HCC recurrence confirmed by imaging.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 3 years
  The overall survival (OS) was defined as the period between the day of LT and the day of the participants' death or the termination of the study in 3 years after LT.

OTHER OUTCOMES:
3-year Recurrence rate (RR) | 3 years
  The 3-year recurrence rate is obtained by dividing the number of recurrence cases in each group by the total number of cases in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Jinyang Gu, PhD, Principal Investigator — Xinhua Hospital Affiliated to Shanghai Jiao Tong University Medical School
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University Medical School, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The IPDs to be shared include study protocol, statistical analysis methods, informed consent form and clinical study report.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available from the manuscript accepted by a journal to five years after that.
Access Criteria: The data will become available when the manuscript accepted by a journal, until five years after that.

REFERENCES:
- [Result] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Result] Briggs A, Daniele B, Dick K, Evans TRJ, Galle PR, Hubner RA, Lopez C, Siebert U, Tremblay G. Covariate-adjusted analysis of the Phase 3 REFLECT study of lenvatinib versus sorafenib in the treatment of unresectable hepatocellular carcinoma. Br J Cancer. 2020 Jun;122(12):1754-1759. doi: 10.1038/s41416-020-0817-7. Epub 2020 Apr 8. PMID 32265508
- [Result] Siegel AB, El-Khoueiry AB, Finn RS, Guthrie KA, Goyal A, Venook AP, Blanke CD, Verna EC, Dove L, Emond J, Kato T, Samstein B, Busuttil R, Remotti H, Coffey A, Brown RS Jr. Phase I trial of sorafenib following liver transplantation in patients with high-risk hepatocellular carcinoma. Liver Cancer. 2015 Mar;4(2):115-25. doi: 10.1159/000367734. PMID 26020033
- [Result] Teng CL, Hwang WL, Chen YJ, Chang KH, Cheng SB. Sorafenib for hepatocellular carcinoma patients beyond Milan criteria after orthotopic liver transplantation: a case control study. World J Surg Oncol. 2012 Feb 17;10:41. doi: 10.1186/1477-7819-10-41. PMID 22339891